CLINICAL TRIAL: NCT00156273
Title: A Pilot Study to Determine the Feasibility of Quantifying Apoptosis and Bcl-2 Expression in Circulating Tumor Cells (CTCs) in Women Undergoing Treatment for Metastatic Breast Cancer
Brief Title: Determine Feasibility of Quantifying Apoptosis and Bcl-2 Expression in CTCs in Women With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2003.075; HUM 45808 Legacy 2004-0703 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We are trying to develop better ways to detect when cancer therapies are working.

ELIGIBILITY:
Inclusion Criteria:

1.Females at least 18 years of age 2 Diagnosis of metastatic breast cancer 3.ECOG Score of 0-2 4.Treating oncologist has decided to initiate any new systemic therapy with emphasis on recruiting patients commencing a taxane-based regimen. Taxine-based therapy may be docetaxel or paclitaxel, and it can be given on any schedule,including weekly or every 3 weeks. Other treatment can include non-taxane chemotherapy or trastuzumab-with or without other therapy.

5.Patient is willing to return for one or more additional ~18 mL blood draw (s) at 24-48-, and /or 72 hours and ~3-4 weeks after the initiation of therapy.At a minimum, patients must donate blood at baseline, one intermediate interval (24, 48, 72 hr) and at ~3-4 weeks 6.Signed Informed Consent Form

-

Exclusion Criteria:

Patient is unable and unwilling to provide a blood specimen at a minimum of one of the intermediate blood draw time points at 24, 48, or 72 hours -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2005-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of detecting Bcl2 expression and apoptosis in CTCs | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Smerage, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States